CLINICAL TRIAL: NCT07056270
Title: Development of a Set of Auxiliary Decision-making System for the Perioperative Period of Hepatectomy Based on Static CT and Artificial Intelligence.
Status: Not yet recruiting | Type: Observational
Sponsor: Tongji Hospital (Other)
Collaborators: Suzhou Institute of Biomedical Engineering and Technology of the Chinese Academy of Sciences (Unknown)
Responsible Party: Principal Investigator, Chen Xiaoping, Chairman of the Department of Surgery, Tongji Hospital
Other Study IDs: CTLIVERai
Record Dates: First submitted 2025-06-29; First posted 2025-07-09 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-06

CONDITIONS: Liver Cirrhosis; Liver Cancer
Keywords: liver cancer; liver cirrhosis; liver resection; microvascular invasion; liver function; static CT
MeSH Terms: conditions — Liver Cirrhosis; Liver Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Biospecimen Retention: Samples Without DNA — Surgical resection specimens of liver cancer
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Static CT group: Patients with chronic liver disease and liver cancer receive static CT scans
  Interventions: Other: static CT scans

INTERVENTIONS:
Other: static CT scans — Patients with chronic liver disease and liver cancer received static CT scans before hepatectomy to establish a high-definition CT database.

SUMMARY:
The study will prospectively recruit patients with chronic liver disease and liver cancer for static CT scans to establish a high-definition CT database. Combining clinical data and pathological information, artificial intelligence technology will be utilized to construct models for assessing liver function and liver cirrhosis, as well as predicting microvascular invasion (MVI).

DETAILED DESCRIPTION:
Liver cancer is a common disease that seriously endangers public health in China, and CT technology is particularly critical in the diagnosis and treatment of liver cancer. Most patients with liver cancer in China are complicated with liver cirrhosis, and the treatment principle is a comprehensive model based on surgical resection. The main problem in the perioperative period of hepatectomy is to accurately evaluate the grade of cirrhosis, liver reserve function and predict microvascular invasion (MVI) before operation. In view of these problems, this project plans to develop a set of auxiliary decision-making system for the perioperative period of hepatectomy of liver cancer based on static CT and artificial intelligence technology and combined with expert consensus. The system will first establish a set of high-quality liver health/disease image database based on static CT (slice thickness 0.165mm, 2048×2048 scanning/reconstruction matrix, multi-energy spectrum), providing high-quality data source for clinical application development; Then, use artificial intelligence technology to optimize the output high-quality data, data mining and learning, and carry out targeted analysis from the aspects of liver cirrhosis grading, liver reserve function and MVI evaluation; Finally, on the basis of evidence-based medicine and expert consensus, intelligently fuse the multimodal biomedical information to form a set of auxiliary decision-making system for the perioperative period of hepatectomy for liver cancer, which provides a new method for further standardizing the diagnosis and treatment behavior of liver cancer and improving the surgical treatment effect of liver cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are clinically diagnosed with primary liver cancer and other space-occupying liver lesions preoperatively and are planned for surgical resection, or those with underlying liver diseases and cirrhosis;
2. Aged 18-75 years;
3. Willing to participate in this study and have signed the informed consent.

Exclusion Criteria:

1. Planned or unplanned pregnancy and pregnant women;
2. Glomerular filtration rate (GFR) ≤60 ml/min;
3. History of contrast media allergy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are clinically diagnosed with primary liver cancer and other space-occupying liver lesions preoperatively and are planned for surgical resection, or those with underlying liver diseases and cirrhosis
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2027-08 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
microvascular invasion | 7 days after surgery
  microvascular invasion based on pathology
liver cirhosis | 7 days after surgery
  liver cirhosis according to laennec grading system
liver function | 1 day before static CT scanning
  liver funcion based Child-Pugh grading system

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoping Chen, M.D., Study Director — Hepatic Surgery Center, Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not to be shared to protect patient privacy.